CLINICAL TRIAL: NCT03598764
Title: Feasibility and Outcomes of External Pop-out Versus Classic Fetal Head Extract During Cesarean Section: A Randomized Clinical Trial
Brief Title: External Pop-out and Classic Fetal Head Extract During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPCS
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic head extraction group (Other)
  Interventions: Procedure: Classic head extraction during Cesarean section
- External Pop out group (Other)
  Interventions: Procedure: External pop out technique

INTERVENTIONS:
Procedure: Classic head extraction during Cesarean section — by putting the fingers of the right inside the lower uterine segment to deliver the head
  Arms: Classic head extraction group
Procedure: External pop out technique — The palmar aspect of the fingers will be resting on the uterovesical peritoneal reflection not directly on the fetal head.
  Arms: External Pop out group

SUMMARY:
Cesarean section is the delivery of the fetus through a surgical incision in the abdominal wall (laparotomy) and uterine wall (hysterotomy). The rate of cesarean delivery has increased progressively in the last decades until it becomes the most common operation performed all over the world.

A multitude of efforts had been done aiming at a reduction of cesarean section related maternal morbidities; most of them are related to technical modifications of how to open and how to close the abdominal and uterine incisions. The comparative studies of blunt versus sharp extension of the uterine incision showed a reduction of the incidence of unintended extension from 8.8% to 4.8%.

Delivery of the fetal head through the uterine incision is one of the major technical problems during elective cesarean section, especially when the presenting part is non-engaged. All of the previously described procedures, alternative to the classic manual head extraction, were inconclusive and not convincing to the obstetricians for routine use.

Also, no reported well-designed trials favor one of them over other. Application of vacuum cup, use of forceps blade, increasing fundal pressure and making additional uterine incisions were previously reported as alternative techniques. None of them gain any popularity or proved to be used as a basic step during cesarean section, besides many complications were reported due to their use on mothers and infants.

The vulnerability of the lower uterine segment for tears is related to the stage of labor. The frequency of unintended extension was reported to be 15.5%, and 35.0% in cases operated in first and second stages of labor respectively.

As with any surgical operation, anticipating difficulties during cesarean delivery and avoiding these difficulties is always the greatest practice. Although much has been written about techniques for managing difficult head extraction during vaginal deliveries, the reports addressed the management of difficult head delivery during cesarean section in literature are scarce.

The original techniques of fetal head extraction entail the introduction of the obstetricians hand or other instruments into the lower uterine segment. This puts the lower uterine segment at risk of damage and incision extensions with its consequences of increased blood loss, increased operative time, infection, adhesion and blood transfusion. Adherence to the available the generated good quality evidence bases practice in cesarean section is anticipated to decrease such morbidities.

The idea of the present technique was derived from the fact that during vaginal delivery the main task of the obstetrician is to support the perineum while the fetal head extends to get out through birth canal.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women in single, living, term (>37 weeks), cephalic fetus.
2. Women eligible for elective Cesarean section.

Exclusion Criteria:

1. Multiple gestations
2. Placenta previa
3. Fetal congenital anomalies as hydrocephalus
4. Intrauterine fetal death.
5. US evidence anhydramnios

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 910 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Number of women developed uterine tears | 5 minute

SECONDARY OUTCOMES:
Time of head extraction (minutes) | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No